CLINICAL TRIAL: NCT04673318
Title: Physical Rehabilitation of COVID-19 Survivors by Heat Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2151
Record Dates: First submitted 2020-10-23; First posted 2020-12-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Physical Disability
Keywords: physical rehabilitation; cardio-vascular function; metabolism; heat therapy
MeSH Terms: conditions — COVID-19; Hyperthermia | interventions — Diathermy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Course of recovery with standard of care.
- Exercise training (Active Comparator): low resistance velocity based exercise training ~40 min, 3 times a week at home for 8 weeks
  Interventions: Behavioral: exercise training
- heat therapy (Experimental): heat therapy (~40C skin temperature) with a leg garment 5 times a week for 40-55 min for 8 weeks
  Interventions: Behavioral: heat therapy

INTERVENTIONS:
Behavioral: heat therapy — leg heated garments with circulating water to conduct heat therapy at home
  Other Names: exercise training
  Arms: heat therapy
Behavioral: exercise training — A velocity based training program will be implemented at home using a mobile app allowing for the quantification the relative intensity.
  Arms: Exercise training

SUMMARY:
Older adults and people with underlying medical conditions are at higher risk for developing serious complications related to SARS-CoV-2 resulting in prolonged sequelae. The goal of this proposal is to compare the benefits of home-based lower limb heat therapy to exercise training on cardio-metabolic function and mobility in older adults during their convalescence from hospitalization due to SARS-CoV-2.

DETAILED DESCRIPTION:
The novel coronavirus (severe acute respiratory syndrome [SARS]-CoV-2), first identified in December 2019 in Wuhan, China, has since spread worldwide. Older adults and people with underlying medical conditions are at higher risk for developing serious complications and death related to SARS-CoV-2. However, another challenge is arising in regards to the long-term prognosis of COVID-19 survivors. Although limited, the available data on the medium-term outcomes of patients who survived COVID-19 all indicate prolonged symptom duration and disability in a large proportion of adults hospitalized with severe symptoms. In addition, these patients, a majority of whom were older adults or patients with pre-existing health conditions, spent ~10-15 days bedridden and under intensive treatment, which can have lasting consequences on metabolism and cardiovascular functions, mobility, and eventually lead to long-term disabilities. Upon discharge from the hospital, the main option for physical rehabilitation involves exercise training. Although, exercise training can be effective to restore physical function, it is oftentimes associated with low adherence. Considering the severe deconditioning accompanying hospitalization related to COVID-19, there is a critical need for the development of a rehabilitation strategy that is home-based and practical to individuals with diminished physical function. Accordingly, the goal of this project is to compare the benefits of home-based lower limb chronic heat therapy to exercise training on skeletal muscle metabolism, vascular function and functional capacity in older adults during their convalescence from hospitalization due to SARS-CoV-2. Late middle-age and older adults that have been discharged from a COVID-19 hospitalization will be randomly allocated to an exercise intervention group (EX, low resistance ~40 min, 3 times a week at home), a heat-treated group (HT, leg heated garments with skin temperature reaching ~40˚C, 40-55 min, 5 times a week at home), or a control group (CT) for 8 weeks. Specific Aim 1 will test the hypothesis that local heat therapy in previously hospitalized COVID-19 patients can (i) enhance functional capacity, resulting in improvements in mobility and quality of life compared to a non-treated control group, and (ii) that these changes will be similar in magnitude to an exercise intervention. Specific Aim 2 will test the hypothesis that local heat therapy in the same patients can (i) enhance insulin sensitivity as a consequence of improvements in mitochondrial and vascular function compared to a non-treated control group, and (ii) that these changes will be similar in magnitude to an exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women must not be taking hormone therapy
* Must have been hospitalized for, at least, 5 days for a COVID-19 related infection
* Must have been discharged from the hospital for, at least, 14 days

Exclusion Criteria:

* Orthopedic limitations that would prohibit from performing plantar-flexion or knee-extension exercise
* Contraindication to MRI (pacemaker, metal implants, or certain types of heart valves), or be at medical risk from undergoing an MRI examination
* Enrolled in a rehabilitation program
* BMI <40 kg/m2 and weigh <400lbs
* prior history of pulmonary embolism or deep vein thrombosis

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 8 weeks
  6-min walking distance

SECONDARY OUTCOMES:
Motor function | 8 weeks
  Short Physical Performance Battery score
Glucose control | 8 weeks
  insulin and glucose levels during oral glucose tolerance test
Skeletal muscle mitochondrial function | 8 weeks
  Change in phosphocreatine recovery kinetics measured by 31-PMRS
Vascular function | 8 weeks
  Change in reactive hyperemia

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Applied Life Sciences, Amherst, Massachusetts, United States